CLINICAL TRIAL: NCT02630667
Title: The Acute Effects of Fortified Nutritional Supplementation on Cognition, Memory, & Achievement
Brief Title: The Acute Effects Fortified Nutritional Supplementation on Childhood Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 12641
Record Dates: First submitted 2015-08-25; First posted 2015-12-15 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Cognitive Ability, General; Dietary Modification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SLOW Carbohydrate (Experimental): Treatment consists of a carbohydrate blend designed to elicit a slow postprandial glycemic response.
  Interventions: Other: SLOW Carbohydrate
- MEDIUM Carbohydrate (Experimental): Treatment consists of only one carbohydrate source designed to elicit a medium/moderate postprandial glycemic response.
  Interventions: Other: MEDIUM Carbohydrate
- FAST Carbohydrate (Experimental): Treatment consists of only one carbohydrate source designed to elicit a fast postprandial glycemic response.
  Interventions: Other: FAST Carbohydrate
- Non-Caloric Placebo (Placebo Comparator): Non-caloric placebo consisting of artificial sweeteners
  Interventions: Other: SLOW Carbohydrate; Other: MEDIUM Carbohydrate; Other: FAST Carbohydrate

INTERVENTIONS:
Other: SLOW Carbohydrate — Treatment consists of a carbohydrate blend designed to elicit a slow postprandial glycemic response
  Arms: Non-Caloric Placebo; SLOW Carbohydrate
Other: MEDIUM Carbohydrate — Treatment consists of only one carbohydrate source designed to elicit a medium/moderate postprandial glycemic response
  Arms: MEDIUM Carbohydrate; Non-Caloric Placebo
Other: FAST Carbohydrate — Treatment consists of only one carbohydrate source designed to elicit a fast postprandial glycemic response
  Arms: FAST Carbohydrate; Non-Caloric Placebo

SUMMARY:
The aim of this study is to investigate the acute effects of ingestion of carbohydrates - with different glycemic profiles - on cognitive function among preadolescent children (i.e., 9-10 years).

DETAILED DESCRIPTION:
Regular breakfast consumption is linked to improved cognitive performance in school-aged children. However, the acute benefits of defined nutrient consumption on brain and cognitive health are not well understood, particularly in preadolescent children. One factor that may relate to brain health and learning in children is the contribution of carbohydrates to the digestion rate of a meal (and associated effects on post-prandial glycemia).

The effects of differentially absorbed carbohydrates on brain and cognition are unknown, especially when ingested via a fortified nutritional beverage providing a balanced array of nutrients. The aim of this study is to investigate the acute, transient effect of nutrient supplementation with varied carbohydrate systems in preadolescent children (i.e., 9-10 years).

Participants will be randomized to receive one of three treatment nutritional formulations containing carbohydrates with varying absorption rates along with a non-caloric placebo. Participants will perform a cognitive battery in the fasted condition, shortly after treatment ingestion, and an hour after ingestion. Group differences in performance will be contrasted to assess the effects of different carbohydrate types on children's cognitive function following an overnight fast.

Findings from this study will inform our understanding of the macronutrient profile of breakfast that may potentially improve children's cognitive performance in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Parental/guardian consent.
* Participants must be between the ages of 9-10 years old at the time of testing age
* Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive task (below 20/20 vision).
* Participants must have an IQ > 85 (IQ < 85).

Exclusion Criteria:

* Prior diagnosis of cognitive or physical disability, including ADHD (severe asthma, epilepsy, and dependence upon a wheelchair/walking aid, and ADHD Rating Scale score below 85%).
* Use of anti-psychotic, anti-depressant, anti-anxiety medication, as well as those medications used for ADD/ADHD (use of any anti-psychotic, anti-depressant, anti-anxiety, and ADD/ADHD medications).
* Early pubertal status, as measured by a modified test of the Tanner Staging System (onset of puberty as determined by Tanner).
* Lactose intolerance
* Allergies to milk and/or soy
* Adherence to a strict vegan diet

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2012-06; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Control at 15 minutes Postprandial | 15 minutes Postprandial
  Performance will be assessed using the difference in inverse efficiency (during a modified flanker task) between performance at 15 minutes and baseline/fasted (within 2 hours of wake-time) performance.
Change in Cognitive Control at 70 minutes Postprandial | 70 minutes Postprandial
  Performance will be assessed using the difference in inverse efficiency (during a modified flanker task) between performance at 70 minutes and baseline/fasted (within 2 hours of wake-time).

SECONDARY OUTCOMES:
Change in Relational Memory at 30 minutes Postprandial | 30 minutes Postprandial
  Performance will be assessed using the difference in number of swap errors (during a spatial reconstruction task) by calculating the difference between number of errors performed at baseline/fasted (within 2 hours of wake-time) from number of errors at 30 minutes postprandial.
Change in Relational Memory at 85 minutes Postprandial | 85 minutes Postprandial
  Performance will be assessed using the difference in number of swap errors (during a spatial reconstruction task) by calculating the difference between number of errors performed at baseline/fasted (within 2 hours of wake-time) from number of errors at 85 minutes postprandial.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hillman, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Department of Kinesiology and Community Health, Urbana, Illinois, United States

REFERENCES:
- [Derived] Walk AM, Raine LB, Kramer AF, Cohen NJ, Hillman CH, Khan NA. Adiposity is related to neuroelectric indices of motor response preparation in preadolescent children. Int J Psychophysiol. 2020 Jan;147:176-183. doi: 10.1016/j.ijpsycho.2019.10.014. Epub 2019 Nov 19. PMID 31756405